CLINICAL TRIAL: NCT01118728
Title: A Multicenter Uncontrolled Extension Study Evaluating the Long Term Safety and Efficacy of SAR153191 in Patients With Ankylosing Spondylitis (AS)
Brief Title: Extension Study for Long Term Evaluation of SAR153191 (REGN88) in Patients With Ankylosing Spondylitis
Acronym: SUSTAIN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of benefit on efficacy
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS11298; 2010-019263-11 (EudraCT Number)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sarilumab (Experimental): Sarilumab 150 mg subcutaneous (SC) injection every week (or every other week in case of safety issue) for 260 weeks, or until commercially available, or until discontinuation of the project, whichever came first.
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: SAR153191; REGN88

SUMMARY:
Primary Objective:

* To assess the long term safety of Sarilumab (SAR153191/REGN88) in participants with ankylosing spondylitis (AS)

Secondary Objective:

* To assess the long term efficacy of Sarilumab (SAR153191/REGN88) in participants with AS

DETAILED DESCRIPTION:
The maximum study duration per participant was to be 267 weeks (approximately 5 years) broken down as follows:

* screening up to a maximum of 1 week;
* treatment up to a maximum of 260 weeks;
* follow-up of 6 weeks after treatment discontinuation.

ELIGIBILITY:
Inclusion criteria:

* Participant with AS who participated and completed 12-week treatment in study DRI11073-NCT01061723.

Exclusion criteria:

* Adverse event(s) having lead to treatment discontinuation in the DRI11073 study;
* Event or laboratory abnormality observed at the last treatment visit of DRI11073 study that would have adversely affected participation of the participant in this study as per investigator judgment.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 56 centers in 12 countries. A total of 224 participants were screened between 01 June 2010 and 03 June 2011.
Pre-assignment Details: Of 224 screened participants, 223 participants were enrolled and treated. One participant withdrew consent before randomization.
Period: Overall Study
Arm/Group | Sarilumab
Started | 223
Completed | 0
Not Completed | 223
Not completed — Adverse Event | 17
Not completed — Lack of Efficacy | 27
Not completed — Sponsor's decision to discontinue study | 172
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of the study treatment after signature of the informed consent.
Groups:
- Sarilumab: Sarilumab 150 mg SC injection every week (or every other week in case of safety issue) for 260 weeks, or until commercially available, or until discontinuation of the project, whichever came first.
Arm/Group | Sarilumab
Number analyzed (Participants) | 223
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Treatment-emergent Adverse Event (TEAE), Serious Adverse Event (SAE) and Treatment Discontinuation
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of the relationship to the investigational medicinal product (IMP). SAE was any untoward medical occurrence that at any dose resulted in death or was life-threatening or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect or was a medically important event. TEAEs were AEs that developed or worsened or became serious during the TEAE period (time from first dose of IMP up to the end of follow-up period).
Time Frame: Baseline up to the end of study (66 weeks)
Population: Analysis was performed on safety population defined as all participants who received at least one dose of the study treatment after signature of the informed consent.
Measure: Number; unit: Percentage of participants
Arm/Group | Sarilumab
Number analyzed (Participants) | 223
Percentage of participants
  Any TEAE | 67.3
  Any treatment-emergent SAE | 5.4
  Any TEAE leading to treatment discontinuation | 8.1

2. Secondary Outcome: Percentage of Participants Who Achieved 20% Response in Ankylosing Spondylitis (AS) Working Group Criteria for Response (ASAS20)
Description: Treatment response for ASAS20 was defined as: Improvement of ≥ 20% and ≥ 1 unit on a 0 (least) to 10 (worst) numerical rating score (NRS) in at least 3 of the 4 ASAS improvement criteria (ASASIC) domains, and no worsening of ≥ 20% and ≥ 1 unit on 0-10 NRS in the remaining domain. The 4 domains included were participant's global disease activity assessment, total back pain, physical function (Bath Ankylosing Spondylitis Functional Index), and Inflammation (mean of last 2 Bath Ankylosing Spondylitis Disease Activity Index questions on morning stiffness).
Time Frame: Baseline up to the end of treatment (60 weeks)
Population: Analysis was performed on safety population. Number of participants analyzed=participants with ASAS20 assessment at specified time-points. Here 'n' signifies number of participants with available data for specified time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | Sarilumab
Number analyzed (Participants) | 218
Percentage of participants
  Week 0 (n=218) | 30.3
  Week 12 (n=207) | 40.1
  Week 24 (n=150) | 46.0
  Week 36 (n=93) | 41.9
  Week 48 (n=37) | 59.5
  Week 60 (n=7) | 57.1

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to the final visit (Day 414) regardless of seriousness or relationship to investigational product
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from first dose of IMP up to the end of follow-up period).
Arm/Group | Sarilumab
Serious Adverse Events (participants affected / at risk) | 12/223
Other Adverse Events (participants affected / at risk) | 62/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab (N=223)
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Tuberculin test positive (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab (N=223)
Nasopharyngitis (Infections and infestations) | 16
Upper respiratory tract infection (Infections and infestations) | 13
Neutropenia (Blood and lymphatic system disorders) | 21
Aphthous stomatitis (Gastrointestinal disorders) | 12
Injection site reaction (General disorders) | 14

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued after approximately 1.5 years, when the ankylosing spondylitis development program was discontinued due to lack of efficacy in the DRI11073 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.